CLINICAL TRIAL: NCT06930820
Title: In-Hospital Electronic Registry of Severe Trauma of the Fondazione I.R.C.C.S. Policlinico San Matteo (TRAUMA REGISTRY S. MATTEO)
Brief Title: In-Hospital Electronic Registry of Severe Trauma of the Fondazione I.R.C.C.S. Policlinico San Matteo
Acronym: STRAP register
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Luca Ansaloni, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: S.Matteo TRAuma Pavia Registry
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-02

CONDITIONS: Patients Who Are Victims of Major Trauma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The objective of establishing an in-hospital Trauma Registry, aimed at collecting data on patients who are victims of major trauma and treated at our Center, is to develop a comprehensive and in-depth tool for the analysis and monitoring of clinical activity within a Level I Trauma Center. The purpose of building such databases-specifically the proposed Trauma Registry-is to provide the hospital with a unique instrument for analyzing and monitoring the epidemiology and management of a specific patient population.

In light of recent developments in the hospital's newly implemented clinical care pathway (PDTA) for the management of polytrauma patients, and the strategic enhancement offered by the opening of a dedicated helipad for the reception of such patients, our working group is committed to promoting a tool that may, both in the short and long term, foster clinical and scientific advancement at the Fondazione I.R.C.C.S. Policlinico San Matteo in Pavia.

Our general objective is the prospective collection of data on major trauma patients admitted to and treated at the Fondazione I.R.C.C.S. Policlinico San Matteo.

Our primary objective is to evaluate in-hospital mortality, used as a qualitative indicator of the Trauma Center's performance, among patients with severe trauma managed at our institution.

ELIGIBILITY:
Inclusion Criteria:

All consecutive patients presenting to the Emergency Department of the Fondazione I.R.C.C.S. Policlinico San Matteo who meet at least one of the following criteria will be included in the registry:

* They were transported to the Emergency Department by Emergency Medical Services (AREU - Regional Emergency and Urgency Agency) with a diagnosis of Severe Trauma / Major Trauma

or

- They arrived at the Emergency Department and were admitted with a diagnosis of "trauma", and were found, upon completion of the secondary assessment, to have an Injury Severity Score (ISS) >15

Exclusion Criteria:

There are no exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are victims of major trauma
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2032-07-07 (Estimated); Study Completion 2032-07-07 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality rate | through study completion, an average of 10 years
  The primary objective of the registry is to evaluate in-hospital mortality for patients with severe trauma treated at the Fondazione I.R.C.C.S. Policlinico San Matteo.

SECONDARY OUTCOMES:
Relationship between the severity of traumatic injuries, quantified using the Injury Severity Score (ISS), and in-hospital mortality | through study completion, an average of 10 years
  Evaluation of the relationship between the severity of traumatic injuries, quantified using the Injury Severity Score (ISS), and in-hospital mortality.
Hospital length of stay and its relationship with the ISS | through study completion, an average of 10 years
  Evaluation of hospital length of stay and its relationship with the ISS.
Intensive Care Unit (ICU) length of stay and its relationship with the ISS | through study completion, an average of 10 years
  Evaluation of Intensive Care Unit (ICU) length of stay and its relationship with the ISS.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Pavia, Italy